CLINICAL TRIAL: NCT07317973
Title: Patient Decision Aids for Childhood Type 1 Diabetes Screening, Follow-Up, and Enrolment in Trials
Brief Title: A Study About Patient Decision Aids Designed to Help Parents and Guardians in Canada Make Evidence-informed, Values-congruent Decisions About Screening Children for Type 1 Diabetes and Follow-up Decisions.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: CanScreenT1D PtDAs
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-10

CONDITIONS: Diabetes, Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient decision aid (Experimental): Participants receive patient decision aid
  Interventions: Other: Web-based patient decision aid
- Control (Active Comparator): Participants receive standard materials
  Interventions: Other: Standard materials

INTERVENTIONS:
Other: Web-based patient decision aid — The web-based patient decision aid will provide information and support decisions relevant to screening children for type 1 diabetes and follow-up according to screening results.
  Arms: Patient decision aid
Other: Standard materials — Standard materials provided to parents whose children are eligible for type 1 diabetes screening and follow-up.
  Arms: Control

SUMMARY:
This study will design and test patient decision aids to help parents and guardians in Canada make decisions about screening their children for type 1 diabetes. To do this, we will work with a panel of parents and guardians as well as scientific experts, show draft designs to parents and guardians, improve the draft designs based on feedback, and finally test the patient decision aids in online studies.

DETAILED DESCRIPTION:
BACKGROUND: A new consortium funded by Breakthrough T1D Canada (formerly Juvenile Diabetes Research Foundation Canada) and the Canadian Institutes of Health Research (CIHR) is exploring childhood screening for risk of type 1 diabetes (T1D) in the general population in Canada. Childhood screening requires decision making on the part of parents and guardians.

OBJECTIVE: The aim of this study is to develop patient decision aids to support Canadian families facing T1D screening and monitoring-related decisions (whether to screen their children for T1D using genetic or antibody testing, whether to participate in trials investigating medicines to delay or prevent the onset of T1D) by co-designing, optimizing, and evaluating patient decision aids. Patient decision aids are structured tools-often in the form of websites or pamphlets-intended to complement and support shared decision making with health care professionals. They specifically support decision making by making the decision explicit, providing information on potential benefits and harms of each option, and helping people clarify what matters most to them pertaining to the decision.

METHODS: We will work with an advisory committee of parents and guardians from across Canada and with diverse backgrounds and perspectives to design the patient decision aids. We will then conduct user testing across Canada with both remote and in-person user testing options. Finally, we will conduct online randomized controlled trials of the final patient decision aids to ascertain their effects on measures of decision quality compared to standard materials.

RESULTS: We will assess five measures of decision quality: knowledge, decisional conflict, risk perceptions, decision intentions, and values congruence.

CONCLUSIONS: This project will deliver optimized, evidence-based patient decision aids designed to support Canadian families (i.e., parents/guardians) in making informed, values-congruent decisions about T1D screening, follow-up, and enrollment in clinical trials for their child(ren). Our final audience for this work will be parents and guardians across Canada. We plan to offer the patient decision aids in the screening program pilot study and eventually scale up dissemination of the decision aids through registration in a known decision aid repository (decisionaid.ohri.ca) and collaborations with public health agencies of participating provinces. We will seek inclusion in online patient portals where such options exist.

ELIGIBILITY:
Inclusion Criteria:

Participants must be 18 or older, live in Canada, be able to read and understand either English or French, and be able to use a computer. They must not have uncorrected visual and/or hearing impairments, currently have one or more children and be eligible to make a decision about T1D screening for a current (already born) or future (currently expected due to pregnancy) child.

Exclusion Criteria:

All participants who do not complete the visualization of the tools for various reasons (lack of availability, strong emotions, internet connection problems, etc.) will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Knowledge | Immediately post-intervention
  To assess knowledge, we will develop a questionnaire specific to the topic of screening for T1D based on previous work by the developers of the Ottawa Decision Support Framework [https://decisionaid.ohri.ca/eval_know.html] and building on work conducted by members of the CanScreenT1D consortium to develop a core outcomes set relevant to T1D screening. [https://doi.org/10.1136/bmjopen-2025-099537] Answers to each question will receive a score of 1 (if the participant selects the correct answer "true" or "false") and 0 (if the answer is incorrect or if the participant answers "uncertain"). Items are totaled and an average knowledge score is calculated. For comparison with scales from 0 to 100, the score can be converted into a percentage of correct answers.
Decisional conflict | Immediately post-intervention
  To assess decisional conflict, we will use the validated 16-item Decisional Conflict scale. [https://doi.org/10.1177/0272989X9501500105] This scale measures personal perceptions of a) uncertainty in the choice of options; b) modifiable factors contributing to uncertainty, such as feelings of being uninformed, unclear about personal values and unsupported in decision-making; and c) decision-making effectiveness, such as feelings that the choice is informed, value-based, actionable and expressions of satisfaction with the choice.

SECONDARY OUTCOMES:
Risk perception | Immediately post-intervention
  Specifically, we will assess risk perception according to measures in the consortium core outcome set. [https://doi.org/10.1136/bmjopen-2025-099537]
Values congruence | Immediately post-intervention
  Values congruence refers to the extent to which a decision aligns with one's personal values. To assess perceived values congruence, we will analyse the Values Clarity subscale of of the Decisional Conflict Scale. [https://doi.org/10.1177/0272989X9501500105] We will also analyse actual congruence between stated values measured prior to the decision on a visual analogue scale with the decision ultimately made.
Decision intentions | Immediately post-intervention
  For decision intentions, we will elicit people's inclination or propensity to choose an option depending on the case (for example, getting one's child a genetic test or antibody tests, or enrolling one's child in follow-up activities such as participation in clinical trials.) We will use a 101-point visual analogue scale with labels at each extremity and in the middle. We will assign a value of -50 to one extremity, with a label such as, "will definitely not get my child tested for antibodies against type 1 diabetes," a value of 0 at the centre with a label such as, "unsure" and a value of +50 at the other extremity with a label such as, "will definitely get my child tested for antibodies against type 1 diabetes."

CONTACTS AND LOCATIONS:
Overall Officials: Holly Witteman, PhD, Principal Investigator — Laval University

IPD SHARING:
Plan to Share IPD: Yes
We plan to share anonymized study data on Laval University's Dataverse (Borealis.)
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: IPD and supporting information will be available following completion of the study and as long as the Borealis instance is available.
Access Criteria: Anyone with internet access will be able to access it.
URL: https://borealisdata.ca/dataverse/laval